CLINICAL TRIAL: NCT02038387
Title: Prospective Clinical Study on the Role of the Immune Response, in Relation to Diet, in Patients With Either Chronic Hepatitis C Virus (HCV) Infection or Non Alcoholic Fatty Liver Disease (NAFLD). Director Prof. V. Barnaba, Head of Internal Medicine; Principal Investigator, Prof. C. Balsano
Brief Title: Prospective Clinical Study of the Role of the Immune Response, in Relation to Diet, in Patients Affected by Either Chronic Hepatitis C Virus (HCV) Infection or Non Alcoholic Fatty Liver Disease (NAFLD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof. Clara Balsano, Prospective clinical study on the role of the immune response, in relation to diet, in patients affected by either chronic hepatitis C virus (HCV) infection or non alcoholic fatty liver disease (NAFLD), University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 717/12
Record Dates: First submitted 2013-12-13; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Hepatitis C Virus; Non Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Hepatitis C, Chronic; Non-alcoholic Fatty Liver Disease

ARMS (1):
- Diet (Experimental)
  Interventions: Behavioral: normocaloric low cholesterol diet

INTERVENTIONS:
Behavioral: normocaloric low cholesterol diet

SUMMARY:
Chronic hepatitis C virus (HCV) infection and nonalcoholic fatty liver disease (NAFLD) are characterized by a spectrum of pathological conditions ranging from an early stage of inflammation and fibrosis up to more advanced disease conditions, such as hepatocellular carcinoma. The prevalence of NAFLD is between 10 and 25% of the population, with large differences in age and ethnic groups, while it is well known that HCV infection is a major cause of chronic liver disease in Western countries.

For both diseases the progression of liver damage is in close correlation with the lifestyle of patients (eg., nutrition, physical activity, ingestion of alcohol, etc.). In fact, it was shown that feeding imbalances may have implications in altering the normal immune functions of the subjects, suggesting that the metabolic and the immune systems are closely related to each other. Although it is well known the negative role of obesity on the progression of NAFLD and HCV liver diseases, the pathogenic mechanism underlying the alterations related to the immune response is not yet fully understood. Insulin resistance, altered lipid metabolism, lipid peroxidation, oxidative stress and mitochondrial alterations are pathogenic mechanisms that induce liver damage and its progression, both in NAFLD and in HCV infection.

Recent studies suggest that the evolution of viral infections and chronic inflammation in NAFLD are deeply influenced by CD4+ T helper cells expressing IL-17 , defined as T helper 17 (Th17) cells. Broadening the knowledge on the role of diet in the course of NAFLD and HCV infection in the activation of Th17 cells and in the alteration of some of their functions, will allow to shed light on the pathogenic mechanisms underlying the progression of immune-mediated diseases. Moreover, this investigation will allow to understand whether Th17 cells may have a role in the diminished response to therapy in patients who have high cholesterol levels.

If the results will confirm our hypothesis, this study will provide useful informations for the clinical management of patients with both steatosis and chronic HCV infection. The data obtained can also be used for the development of new therapeutic strategies directed to modulate the antiviral immune response.

All patients will undergo clinical and instrumental assessment depending on the type of pathology. Patients will be required to follow a normocaloric low cholesterol diet for a period of 30 days.

The prospective clinical study does not present any form of additional risk for the patients and will be conducted in accordance with the principles established by the Declaration of Helsinki and with the standards of Good Clinical Practice (GCP). The study does not require any additional costs.

ELIGIBILITY:
Inclusion Criteria:

* chronic HCV infection or NAFLD

Exclusion Criteria:

* any pharmacological treatment at least 6 months before entering the study, liver cirrhosis, co-infection by hepatitis B virus, or human immunodeficiency virus infections, autoimmune diseases, and other relevant associated-diseases such as decompensated diabetes, kidney diseases, pulmonary diseases, tumors.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the immune Th17 mediated cell response modulation in subjects with chronic HCV infection vs NAFLD subjects administered with a 30-day low cholesterol diet | Th17 immune response and other liver indices were assessed at baseline and after 30 days of diet. Participants were weekly, up to 4 weeks, followed to assess their adherence.
  Evaluation of the immune Th17 mediated cell response was assessed at baseline and after 30 days by diet administration

CONTACTS AND LOCATIONS:
Overall Officials: Clara Balsano, MD, Study Chair — University of Roma La Sapienza
Locations (1):
- Departemnt of Internal Medicine, La Sapienza University, Rome, Italy

REFERENCES:
- [Derived] Maggio R, Viscomi C, Andreozzi P, D'Ettorre G, Viscogliosi G, Barbaro B, Gori M, Vullo V, Balsano C. Normocaloric low cholesterol diet modulates Th17/Treg balance in patients with chronic hepatitis C virus infection. PLoS One. 2014 Dec 22;9(12):e112346. doi: 10.1371/journal.pone.0112346. eCollection 2014. PMID 25532016